CLINICAL TRIAL: NCT03715972
Title: Cerebrovascular Reserve and White Matter Disease in Patients with Chronic Anemia
Acronym: CVR
Status: Completed | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, John C. Wood, Professor of Pediatrics and Radiology, Children's Hospital Los Angeles
Other Study IDs: CHLA-17-00496; 1R01HL136484-01A1 (NIH)
Record Dates: First submitted 2018-02-20; First posted 2018-10-23 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2023-05

CONDITIONS: Thalassemia; Sickle Cell Disease; Healthy Controls
Keywords: cerebrovascular reserve; white matter disease in patients with chronic anemia
MeSH Terms: conditions — Thalassemia; Anemia, Sickle Cell | interventions — Hydroxyurea; Acetazolamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Anemia Observation: The study will enroll 90 adult subjects with transfusion independent sickle cell disease (70 SS, 10 SC, 10 Sβ0) and 60 patients with transfusion-dependent sickle cell disease. It will also include 10 transfusion independent thalassemia patients and 20 transfusion dependent thalassemia patients. Diamox (acetazolamide) will be administered during MRI.
  Interventions: Drug: Acetazolamide
- Anemia Intervention: Most patients will already be prescribed hydroxyurea as part of their standard of care. Since hydroxyurea could impact brain blood flow, there is also a small pilot study (20 patients, nonrandomized, open label) where MRI imaging will be performed prior to and following administration of hydroxyurea up to maximum tolerated dose.
  non transfusion dependent sickle cell disease patients not already receiving hydroxyurea will be placed on hydroxyurea following their baseline exam and titrated to maximal tolerated dose. They will then undergo a repeat MRI within two months of reaching that dose and be given the option to continue on hydroxyurea or stop.
  Interventions: Drug: Hydroxyurea; Drug: Acetazolamide
- Healthy Controls: 40 control subjects recruited from first degree relatives of the sickle cell disease population. Diamox (acetazolamide) will be administered during MRI.
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Hydroxyurea — info included in arm group
  Other Names: Hydrea
  Groups: Anemia Intervention
Drug: Acetazolamide — Acetazolamide will not be considered a treatment; however, it will be used as a tool to help measure cerebralvascular reserve. A dose of 16 mg/kg ACZ will be administered with a maximum of 1400 mg.
  Other Names: Diamox

SUMMARY:
This is primarily an observational trial in patients with chronic anemia syndromes (sickle cell disease and thalassemia) and control subjects. The key purpose is to understand how brain blood flow reserve (the ability of the brain to increase its flow in response to stress) is altered in patients with chronic anemia. Since this parameter may depend on anemia severity, we will perform the MRI monitoring prior to and following clinically indicated transfusions in a subset of patients. Most patients will already be prescribed hydroxyurea as part of their standard of care. Since hydroxyurea could impact brain blood flow, there is also a small pilot study (20 patients, nonrandomized, open label) where MRI imaging will be performed prior to and following administration of hydroxyurea up to maximum tolerated dose. The study will enroll 90 adult subjects with transfusion independent sickle cell disease (70 SS, 10 SC, 10 Sβ0) and 60 patients with transfusion-dependent sickle cell disease. It will also include 10 transfusion independent thalassemia patients and 20 transfusion dependent thalassemia patients as well as 40 control subjects recruited from first degree relatives of the sickle cell disease population. All eligible subjects will be asked to provide informed consent before participating in the study.

DETAILED DESCRIPTION:
This is primarily an observational trial in patients with chronic anemia syndromes (sickle cell disease and thalassemia) and control subjects. The key purpose is to understand how brain blood flow reserve (the ability of the brain to increase its flow in response to stress) is altered in patients with chronic anemia. Since this parameter may depend on anemia severity, we will perform the MRI monitoring prior to and following clinically indicated transfusions in a subset of patients. Most patients will already be prescribed hydroxyurea as part of their standard of care. Since hydroxyurea could impact brain blood flow, there is also a small pilot study (20 patients, nonrandomized, open label) where MRI imaging will be performed prior to and following administration of hydroxyurea up to maximum tolerated dose. The study will enroll 90 adult subjects with transfusion independent sickle cell disease (70 SS, 10 SC, 10 Sβ0) and 60 patients with transfusion-dependent sickle cell disease. It will also include 10 transfusion independent thalassemia patients and 20 transfusion dependent thalassemia patients as well as 40 control subjects recruited from first degree relatives of the sickle cell disease population. All eligible subjects will be asked to provide informed consent before participating in the study.

Treatment:

All patients will undergo baseline phlebotomy, brain MRI, and neurocognitive testing. The MRI will include measurements of brain blood flow prior to and following administration of 16 mg/kg of acetazolamide to maximally vasodilate the cerebral vasculature. All transfusion dependent patients will have their MRI performed immediately prior to a routinely scheduled transfusion at their hemoglobin nadir. 20 sickle cell disease patients on chronic simple transfusions and 10 thalassemia patients on chronic simple transfusions will undergo repeat MRI assessment of cerebral blood flow and reactivity following their clinically indicated blood transfusion. 10 sickle cell disease patients on exchange transfusions will undergo repeat MRI assessment of cerebral blood flow and reactivity following their clinically indicated exchange transfusion; this transfusion will be performed to lower their hemoglobin S percentage by 25% points while keeping the total hemoglobin unchanged (isocrit exchange). 20 non transfusion dependent sickle cell disease patients not already receiving hydroxyurea will be placed on hydroxyurea following their baseline exam and titrated to maximal tolerated dose. They will then undergo a repeat MRI within two months of reaching that dose and be given the option to continue on hydroxyurea or stop.

Safety Assessment:

All patients will have a physician present during the MRI examination to monitor vital signs and response to acetazolamide. Patients placed onto hydroxyurea will have monthly study visits with monitoring of complete blood count, vital signs, complete metabolic panel, and hemoglobin electrophoresis. Adverse events will be assessed at every study visit after the first dose through to the last subject visit.

Efficacy Assessments:

Baseline cerebrovascular reserve (CVR) predictors will be assessed by multivariate regression after appropriate transformations. Potential independent predictors include oxygen content, hemoglobin subtype, as well as markers of hemolysis, inflammation, and iron overload.

ELIGIBILITY:
* Inclusion Criteria:

  1. Diagnosis of sickle cell disease (genotype SS, SC, or SB0), thalassemia (transfusion dependent or transfusion independent), or normal control subject that are ≥18yrs, ethnicity, and sex matched to the sickle cell disease population.
  2. Ability to tolerate a one hour MRI examination.
  3. Age equal to or greater than 7 years old for Anemia groups.
  4. Agreeable to use an approved method of contraception for the entire duration of hydroxyurea usage if accepted onto the hydroxyurea substudy (male or female of childbearing potential)

Exclusion Criteria:

1. Hospitalization within one month
2. Contraindication to acetazolamide use (seizures)
3. Severe claustrophobia.
4. Pregnancy or nursing (a negative HCG (pregnancy) test must be obtained prior to MRI)
5. As a result of medical review, physical examination or screening investigations, the Principal Investigator (PI) considers the subject unfit for the study
6. No fixed address
7. In control subjects, chronic hepatitis, diabetes, hypertension, coronary artery disease, cognitively impaired or developmental delay

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — for healthy controls we will try to match gender to those that have been enrolled under the anemia cohort
Study Population: sickle cell disease: non-transfused, simple transfused, exchange transfusion Non-sickle Cell Anemia: Non- transfused and transfused healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
CVR response to transfusion | 3-5 days
  Cerebral vascular flow reserve will be assessed prior to and following a regularly scheduled blood transfusion
CVR response to hydroxyurea therapy | 2-4 months
  Change in cerebral vascular reserve at baseline and after initiation of hydroxyurea titrated to maximum tolerated dose

SECONDARY OUTCOMES:
Predictors of CVR response | Single study visit
  We will determine what factors determine cerebral blood flow response to diamox vasodilator challenge

CONTACTS AND LOCATIONS:
Overall Officials: John C Wood, M.D., PhD, Principal Investigator — CHLA/USC
Locations (1):
- CHLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided